CLINICAL TRIAL: NCT01329939
Title: The Effect of Montelukast on Asthma Control in Overweight/Obese Atopic Asthmatics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Thrasher Research Fund (Other); Merck Sharp & Dohme LLC (Industry); New York State Department of Health (Other Government)
Responsible Party: Principal Investigator, Sherry Farzan Kashani, Attending, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-029B
Record Dates: First submitted 2011-03-23; First posted 2011-04-06 (Estimated); Results first posted 2016-04-07 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-03

CONDITIONS: Asthma; Obesity; Inflammation
Keywords: Asthma; Obesity; Pediatric; Inflammation; Leukotriene; Montelukast
MeSH Terms: conditions — Asthma; Obesity; Inflammation | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Obese atopic asthmatics, montelukast (Experimental): Obese/overweight (BMI 85%ile or above for children and > 25 for adults) mild to moderate persistent asthmatics age 7 and above, with environmental allergies who were on daily inhaled corticosteroid treatment and not on montelukast, were randomized to receive montelukast in a double blinded fashion.
  Interventions: Drug: Montelukast
- Lean atopic asthmatics, placebo (Placebo Comparator): Normal weight (BMI less than 85%ile or above for children and < 25 for adults) mild to moderate persistent asthmatics age 7 and above, with environmental allergies who were on daily inhaled corticosteroid treatment and not on montelukast, were randomized to receive placebo in a double blinded fashion.
  Interventions: Drug: Placebo
- Lean atopic asthmatics, montelukast (Active Comparator): Normal weight (BMI less than 85%ile or above for children and < 25 for adults) mild to moderate persistent asthmatics age 7 and above, with environmental allergies who were on daily inhaled corticosteroid treatment and not on montelukast, were randomized to receive montelukast in a double blinded fashion.
  Interventions: Drug: Montelukast
- Obese atopic asthmatics, Placebo (Placebo Comparator): Obese/overweight (BMI 85%ile or above for children and > 25 for adults) mild to moderate persistent asthmatics age 7 and above, with environmental allergies who were on daily inhaled corticosteroid treatment and not on montelukast, were randomized to receive placebo in a double blinded fashion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Montelukast — Age-dependent dose, nightly, 24 weeks
  Other Names: Singulair
  Arms: Lean atopic asthmatics, montelukast
Drug: Placebo — Age-dependent dose, nightly, 24 weeks
  Arms: Lean atopic asthmatics, placebo
Drug: Montelukast — Age-dependent dose, nightly, 24 weeks
  Other Names: Singulair
  Arms: Obese atopic asthmatics, montelukast
Drug: Placebo — Age-dependent dose, nightly, 24 weeks
  Arms: Obese atopic asthmatics, Placebo

SUMMARY:
Background: In recent years, the prevalence of both asthma and obesity has risen dramatically among children and adolescents in the United States. Given the concurrent rise in the two epidemics, there may be an underlying link. Obesity contributes to asthma severity and control, and may play a role in its underlying cause. Obesity is associated with a state of heightened inflammation that may lead to an increase asthma symptoms and severity. Obese adult patients treated with montelukast, an anti-inflammatory agent, seemed to have better asthma control than those treated with other standard asthma medications. The use of montelukast in obese children and adolescents has not been specifically studied.

Hypotheses and Specific Aims: The use of montelukast will improve asthma symptoms and objective markers of asthma to a greater degree in obese, as opposed to non-obese children and adolescents. The investigators would like to determine if the use of montelukast will improve objective asthma scores, pulmonary function, markers of inflammation and medication use to a greater degree in obese as opposed to non-obese children/adolescents.

Potential Impact: Given the growing epidemic of obesity-associated asthma in the U.S., a tailored approach focused on obese asthmatic children may help reduce the burden of this disease, health care costs and potential long-term complications as these children enter adulthood. Furthermore, this study may help clarify the underlying mechanisms that link asthma and obesity. Although this proposal is focused on one medication, it provides an example of how certain medications may have differential efficacy in the obese asthmatic.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate persistent asthma based on 2007 NIH Asthma Guidelines
* age 7-17 years old

Exclusion Criteria:

* present smoking or smoking history
* other significant pulmonary or cardiac condition
* recent (within the past three months) use of montelukast
* on allergen immunotherapy
* on omalizumab
* pregnancy

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2011-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Farzan, MD, Principal Investigator — Northwell Health
Locations (1):
- North Shore-Long Island Jewish Health System, Division of Allergy/Immunology, Great Neck, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Farzan S, Khan S, Elera C, Tsang J, Akerman M, DeVoti J. Effectiveness of montelukast in overweight and obese atopic asthmatics. Ann Allergy Asthma Immunol. 2017 Aug;119(2):189-190. doi: 10.1016/j.anai.2017.05.024. Epub 2017 Jun 28. No abstract available. PMID 28668546

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Atopic asthmatics age seven and above seen in pulmonary and allergy clinics were approached over a 2.5 year period.
Pre-assignment Details: Potential subjects underwent spirometry with bronchodilator administration if there was no previous documentation and allergy testing (skin/blood) to evaluate for environmental allergies.There was a four to six week run-in period where all participants were maintained on an inhaled corticosteroid before randomization.
Groups:
- Overweight/Obese Atopic Asthmatics, Montelukast; Normal Weight Atopic Asthmatics, Montelukast: Montelukast: Age-dependent dose, nightly, 24 weeks
- Normal-weight Atopic Asthmatics, Placebo; Overweight/Obese Atopic Asthmatics, Placebo: Placebo: Age-dependent dose, nightly, 24 weeks
Period: Overall Study
Arm/Group | Overweight/Obese Atopic Asthmatics, Montelukast | Normal-weight Atopic Asthmatics, Placebo | Normal Weight Atopic Asthmatics, Montelukast | Overweight/Obese Atopic Asthmatics, Placebo
Started | 7 | 5 | 5 | 9
Completed | 4 | 4 | 4 | 4
Not Completed | 3 | 1 | 1 | 5
Not completed — Lost to Follow-up | 3 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Obese Atopic Asthmatics, Montelukast | Normal-weight Atopic Asthmatics, Placebo | Normal Weight Atopic Asthmatics, Montelukast | Obese Atopic Asthmatics, Placebo | Total
Number analyzed (Participants) | 7 | 5 | 5 | 9 | 26
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 10 [10 to 15] | 9 [8 to 12] | 10 [9 to 14] | 9 [8 to 16] | 10 [9 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 1 | 6 | 14
  Male | 3 | 2 | 4 | 3 | 12
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 2 | 3 | 2 | 2 | 9
  African-American | 1 | 0 | 1 | 3 | 5
  Hispanic | 0 | 1 | 1 | 2 | 4
  Other | 4 | 1 | 1 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 5 | 9 | 26
Height (cm) [Median (Inter-Quartile Range); unit: cm] | 153.30 [140.4 to 167.64] | 134.4 [132.08 to 139.30] | 143.00 [132.50 to 170.60] | 144.90 [139.7 to 168.00] | 143.95 [134.40 to 167.64]
Weight (kg) [Median (Inter-Quartile Range); unit: kg] | 72.3 [49.30 to 98.88] | 32.66 [27.70 to 34.60] | 37.00 [33.70 to 54.50] | 52.00 [44.20 to 78.00] | 48.50 [36.80 to 73.70]
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 30.76 [22.83 to 34.19] | 17.83 [17.15 to 18.72] | 18.28 [18.09 to 19.20] | 24.20 [22.19 to 27.13] | 22.09 [18.72 to 27.13]

OUTCOME MEASURES:

1. Primary Outcome: Asthma Control Test (ACT) Scores
Description: The ACT is a validated questionaire-based tool designed to assess asthma control. Scale range for 7-11 year olds is 0-27 and for 12 years and older 5-25, with lower scores indicating poorer asthma control for all ages. We did not perform percent change from baseline since in a randomized clinical trial, where the groups are comparable at baseline, we can use only the post-treatment (week 24) data in the analysis.
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Overweight/Obese Atopic Asthmatics, Montelukast | Normal-weight Atopic Asthmatics, Placebo | Normal Weight Atopic Asthmatics, Montelukast | Overweight/Obese Atopic Asthmatics, Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4
units on a scale | 25.00 [22.4 to 27.6] | 20.5 [13.81 to 29.19] | 24.00 [20.10 to 27.90] | 15.75 [3.82 to 27.68]

2. Secondary Outcome: Spirometric Measures
Description: Breathing maneuvers which help to measure obstruction of airways. We did not perform percent change from baseline since in a randomized clinical trial, where the groups are comparable at baseline, we can use only the post-treatment (week 24) data in the analysis.
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: percent predicted
Arm/Group | Overweight/Obese Atopic Asthmatics, Montelukast | Normal-weight Atopic Asthmatics, Placebo | Normal Weight Atopic Asthmatics, Montelukast | Overweight/Obese Atopic Asthmatics, Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4
percent predicted
  FEV1% | 83.37 [66.57 to 100.16] | 85.31 [64.27 to 106.35] | 97.87 [66.55 to 129.19] | 71.79 [47.86 to 95.32]
  FVC% | 91.01 [65.40 to 116.62] | 88.87 [57.89 to 119.85] | 101.68 [69.49 to 133.86] | 76.21 [50.07 to 102.36]
  FEV1/FVC | 83.13 [77.57 to 89.05] | 89.35 [76.38 to 102.31] | 88.25 [75.01 to 101.48] | 80.42 [63.06 to 97.79]
  FEF 25-75% | 87.62 [47.70 to 127.54] | 78.57 [46.25 to 110.88] | 103.77 [49.52 to 158.02] | 66.99 [29.08 to 104.90]
  PEF (peak expiratory flow)% | 100.19 [71.25 to 129.12] | 74.44 [65.05 to 83.84] | 108.09 [74.63 to 141.55] | 92.79 [60.85 to 124.73]

3. Secondary Outcome: Serum Leptin Levels
Description: Leptin levels, measured through blood, mediate appetite and are elaborated by adipose tissue. Levels correlate positively with body fat percentage. In addition, leptin plays a role in producing an inflammatory state. Adiponectin, which is also secreted by adipose tissue, regulates metabolism, however its levels are inversely correlated with body fat percentage.
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Overweight/Obese Atopic Asthmatics, Montelukast | Normal-weight Atopic Asthmatics, Placebo | Normal Weight Atopic Asthmatics, Montelukast | Overweight/Obese Atopic Asthmatics, Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4
ng/mL
  Serum leptin level | 44.35 [29.66 to 59.04] | 4.13 [0.77 to 7.48] | 10.90 [-14.08 to 35.88] | 34.88 [-0.15 to 69.90]
  serum adiponectin | 10.27 [5.66 to 14.88] | 11.35 [0.98 to 21.72] | 13.08 [7.73 to 18.42] | 9.52 [-0.86 to 19.91]

4. Secondary Outcome: Urinary Leukotriene E4 (LTE4) Levels
Description: LTE4 levels, measured in the urine, reflect the degree of inflammation in the asthmatic airway. We did not perform percent change from baseline since in a randomized clinical trial, where the groups are comparable at baseline, we can use only the post-treatment (week 24) data in the analysis.
Time Frame: 24 weeks
Population: One subject in the normal weight atopic asthmatic group who was receiving placebo did not provide a urine sample at 24 weeks.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Overweight/Obese Atopic Asthmatics, Montelukast | Normal-weight Atopic Asthmatics, Placebo | Normal Weight Atopic Asthmatics, Montelukast | Overweight/Obese Atopic Asthmatics, Placebo
Number analyzed (Participants) | 4 | 3 | 4 | 4
pg/mL | 171.50 [39.40 to 303.60] | 195.67 [-460.66 to 852.00] | 198.00 [-80.55 to 476.55] | 313.00 [-227.82 to 853.82]

5. Secondary Outcome: Exhaled Nitric Oxide Measurement
Description: A non-invasive measure of eosinophilic airway inflammation. We did not perform percent change from baseline since in a randomized clinical trial, where the groups are comparable at baseline, we can use only the post-treatment (week 24) data in the analysis.
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: ppb
Arm/Group | Overweight/Obese Atopic Asthmatics, Montelukast | Normal-weight Atopic Asthmatics, Placebo | Normal Weight Atopic Asthmatics, Montelukast | Overweight/Obese Atopic Asthmatics, Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4
ppb | 14.33 [-13.14 to 41.81] | 27.25 [-13.90 to 68.40] | 25.75 [-18.07 to 69.57] | 39.5 [1.7 to 77.2]

6. Secondary Outcome: Beclomethasone Equivalents
Description: The total daily dose of inhaled corticosteroids in beclomethasone equivalents. We did not perform percent change from baseline since in a randomized clinical trial, where the groups are comparable at baseline, we can use only the post-treatment (week 24) data in the analysis.
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: micrograms
Arm/Group | Overweight/Obese Atopic Asthmatics, Montelukast | Normal-weight Atopic Asthmatics, Placebo | Normal Weight Atopic Asthmatics, Montelukast | Overweight/Obese Atopic Asthmatics, Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4
micrograms | 680 [257.80 to 1102.20] | 740 [172.79 to 1652.79] | 580 [302.56 to 857.44] | 1210.00 [456.22 to 1963.78]

7. Secondary Outcome: Urinary Creatinine (Cr) Levels
Description: Creatinine, measured in the urine, reflects how well the kidneys are working, and provide a standard to which one can compare other metabolites in the urine. We did not perform percent change from baseline since in a randomized clinical trial, where the groups are comparable at baseline, we can use only the post-treatment (week 24) data in the analysis.
Time Frame: 24 weeks
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: mg/mL
Arm/Group | Overweight/Obese Atopic Asthmatics, Montelukast | Normal-weight Atopic Asthmatics, Placebo | Normal Weight Atopic Asthmatics, Montelukast | Overweight/Obese Atopic Asthmatics, Placebo
Number analyzed (Participants) | 4 | 3 | 4 | 4
mg/mL | 1.7 [0.95 to 2.45] | 1.69 [-0.36 to 3.75] | 1.77 [-0.18 to 3.73] | 2.77 [0.63 to 4.91]

8. Secondary Outcome: Urinary Creatinine (Cr) Levels/Leukotriene E4 (LTE4) Ratio
Description: The ratio of urinary LTE4 to Cr provides a standardization of the LTE4 level based on the patients weight and muscle mass, therefore normalizing it across the different subjects. We did not perform percent change from baseline since in a randomized clinical trial, where the groups are comparable at baseline, we can use only the post-treatment (week 24) data in the analysis.
Time Frame: 24 weeks
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: pg/mg
Arm/Group | Overweight/Obese Atopic Asthmatics, Montelukast | Normal-weight Atopic Asthmatics, Placebo | Normal Weight Atopic Asthmatics, Montelukast | Overweight/Obese Atopic Asthmatics, Placebo
Number analyzed (Participants) | 4 | 3 | 4 | 4
pg/mg | 105.87 [16.09 to 195.65] | 99.61 [-145.44 to 344.67] | 159.84 [-52.30 to 371.96] | 177.92 [-190.08 to 545.91]

ADVERSE EVENTS:
Arm/Group | Overweight/Obese Atopic Asthmatics, Montelukast | Normal-weight Atopic Asthmatics, Placebo | Normal Weight Atopic Asthmatics, Montelukast | Overweight/Obese Atopic Asthmatics, Placebo
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5 | 0/5 | 0/9
Other Adverse Events (participants affected / at risk) | 0/7 | 0/5 | 0/5 | 3/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overweight/Obese Atopic Asthmatics, Montelukast (N=7) | Normal-weight Atopic Asthmatics, Placebo (N=5) | Normal Weight Atopic Asthmatics, Montelukast (N=5) | Overweight/Obese Atopic Asthmatics, Placebo (N=9)
Mood changes (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"You shall have the right to publish the results derived from your performance of the Study. You agree to submit a copy of...Study results ("Publication") to Merck for comment sixty (60) days prior to its submission for publication. Merck shall have the applicable sixty (60) day period to respond to you with any requested revisions. You agree to delete any confidential information (excluding results) identified by Merck as confidential prior to submitting/presenting the Publication....."